CLINICAL TRIAL: NCT03064802
Title: Multicenter Prospective Registry to Evaluate Use and Outcomes of Burst Biologics Products in Spinal Fusion Surgery
Brief Title: Burst Biologics Spinal Fusion Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Burst Biologics (Industry)
Responsible Party: Sponsor-Investigator, Burst Biologics, Medical Affairs Officer, Smart-Surgical Inc. dba Burst Biologics
Organization: Smart-Surgical Inc. dba Burst Biologics (Industry)
Other Study IDs: SP001
Record Dates: First submitted 2017-02-13; First posted 2017-02-27 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis; Spondylitis; Spondylolisthesis; Herniated Disk
Keywords: BioBurst; Spinal Fusion; Cellular Allograft
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylitis; Spondylolisthesis; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BioBurst Fluid, Burst Allograft: Spinal Fusion with BioBurst Fluid or Burst Allograft
  Interventions: Device: BioBurst Fluid, Burst Allograft

INTERVENTIONS:
Device: BioBurst Fluid, Burst Allograft — BioBurst Fluid or Burst Allograft used to augment spinal fusion

SUMMARY:
A multicenter patient registry was created with aim of documenting how spine and neurosurgeons are utilizing Burst Biologics products along with patient outcomes. These include radiographic measures such as fusion outcome, instrumentation integrity, and clinical outcomes (symptom and function improvement) based on surgeon and patient based outcome assessments.

DETAILED DESCRIPTION:
Spinal fusion surgery remains the most common intervention despite the increasing prevalence of various motion preservation and alternative stabilization devices for patients who are unresponsive to conservative treatment and experience back and/or leg pain and decreased function/quality of life. Donor site morbidity and availability limit the use of autogenous bone and over the past two decades' surgeon interest in alternative bone grafts has steadily increased. Bone morphogenic proteins, synthetic bone graft substitutes, and various allograft products are widely available to surgeons. Limitations on the use of allografts in the past were mainly attributed to less than optimal donor screening and processing techniques which removed viable components needed to aid in the bone healing process.

In recent years, the focus and scientific advances in various allograft processing techniques have allowed the retention of various viable cytokines, growth factors, and cell populations which result in enhanced osteogenic and osteoinductive properties. Rigorous donor bone screening and meticulous testing has virtually eliminated the risk of disease transmission.

A unique proprietary cryoprotection processing technique for allograft tissue was developed by Smart-Surgical, Inc. and a complete line of allograft products was created and is now marketed by Burst Biologics (dba). In addition, rigorous standardized laboratory assay techniques and statistical analysis provide consistency and uniformity of the biologically active components of Burst allograft products.

This prospective registry was designed as an observational study to ascertain how commercially available Burst Products are being used by surgeons performing spinal fusion as well as determining relevant patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient diagnosed with a degenerative spine disorder, has failed conservative treatment, and has decided to undergo surgery.
* The surgeon has determined that a Burst Biologic product is or was clinically indicated.
* Patient capable of understanding the content of the Informed Consent Form
* Patient willing and able to participate in the registry protocol including follow-up visits and clinical evaluations.
* Patient who has agreed to participate in the registry by providing consent according to the applicable local law and the declaration of Helsinki.

Exclusion Criteria:

The following are relative contraindications for the use of Burst Products, however the investigator surgeon is solely responsible for the determination of patient eligibility for surgery:

* Severe vascular or neurological disease
* Uncontrolled diabetes
* Severe degenerative disease (other than degenerative disc disease)
* Hypercalcemia, abnormal calcium metabolism
* Existing acute or chronic infections, especially at the site of the operation
* Inflammatory bone disease such as osteomyelitis
* Malignant tumors
* Patients who are or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the study will be drawn from the individual surgeons practice. Patients will be either candidates for spinal fusion surgery after having failed conservative treatment or will have had spinal fusion surgery and the surgeon determined that the use of a Burst Biologic product is or was clinically indicated.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2017-03-24 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Fusion Rate (%) . Number of patients fused/all patients operated (%) | 12 Months
  Determined by CT Scan or Plain Radiographs

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 12 Months
Change from Baseline in Oswestry Disability Index (ODI) | 12 months
Change from Baseline in Short Form-12 | 12 Months
  SF12 Score
Change from Baseline in Neck Disability Index (NDI) | 12 Months
  NDI Score

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Czop, R.Ph., Study Director — Medical Affairs Officer
Locations (4):
- United States (4):
  - Carrollton Orthopaedic Clinic, Carrollton, Georgia
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - OrthoBethesda, Bethesda, Maryland
  - Cary Orthopedics, Cary, North Carolina

IPD SHARING:
Plan to Share IPD: No